# **Official Title:** Improving Detection and Evidence-based Care of NAFLD in Latinx and Black Patients With Type 2 Diabetes (NAFLD-DM): A Pilot Study

**NCT:** NCT05844137

**IRB Document Date:** 5/31/2024

PI: Anastasia-Stefania Alexopoulos, MD Page **1** of **7** 

Version 2: May 31, 2024

<u>Background</u>: NAFLD is a critically overlooked T2D complication, and T2D accelerates NAFLD progression to poor outcomes, such as cirrhosis, liver cancer and death.<sup>1, 2</sup> As with other T2D complications, **racial and ethnic disparities exist in detection and care of NAFLD**, although the drivers of these disparities are poorly understood, especially in the context of T2D care.<sup>3</sup> Based on my prior work published in *Hepatology*,<sup>4</sup> there are racial/ethnic disparities in who receives liver biopsy to diagnose NAFLD. For instance, of the 350 patients with T2D who underwent liver biopsy for NAFLD between 2007-2019 in DUHS, only 1.7% and 13% of patients were Latinx and Black, respectively.<sup>4</sup> This is striking when considering that these underrepresented minority groups are disproportionately impacted by T2D complications and poor liver outcomes due to NAFLD.<sup>3</sup> Because T2D imparts higher risk of poor liver outcomes due to NAFLD,<sup>1, 2</sup> and because underrepresented minority groups are likewise at higher risk of these outcomes, Latinx and Black patients with T2D should be prioritized for proactive detection and intensive management of NAFLD.<sup>5, 6</sup>

Diabetes care guidelines specifically call for further evaluation of NAFLD in T2D in the presence of abnormal liver enzymes, or when imaging has revealed hepatic steatosis. Detection of high-risk forms of NAFLD is critical in T2D, not only because of the elevated risk of poor NAFLD outcomes in T2D, but also because we can use T2D approaches to effectively treat NAFLD. In a recently published study, we showed that T2D medications that prevent NAFLD progression are vastly underutilized in high-risk patients with T2D. Currently, disparities in the detection and treatment of NAFLD in patients with T2D are poorly characterized; however, given known racial and ethnic disparities in biopsy rates and NAFLD outcomes, we urgently need to understand disparities in NAFLD detection and care in T2D. Such data could directly inform the development of interventions to foster the equitable management of T2D and NAFLD. To address these critical issues, I propose a KL2 program of research that will characterize health disparities in NAFLD detection and care in T2D, and then develop and pilot a culturally-competent intervention that will improve recognition and management of Latinx and Black patients with T2D and NAFLD.

Significance: NAFLD-related liver disease and mortality are high – based on 2015 data, 16.5 million Americans have NASH (i.e., high-risk NAFLD) and mortality in patients with NAFLD is up to 1.27 million annually. These rates are projected to increase by over 130% in the next 10 years. This increased clinical burden will result in direct medical and societal costs of over \$300 billion/year. Efforts to prevent this rise in NAFLD complications and costs should focus on populations at highest risk for poor outcomes; thus, this proposal's focus on T2D and high-risk racial/ethnic groups is highly significant. Furthermore, given known health disparities in NAFLD detection, and in T2D care in general, our emphasis on addressing disparities is crucial. This proposal will generate a patient-facing intervention that will improve evidence-based care of NAFLD in T2D, with a focus on reaching Latinx and Black patients who are disproportionately impacted by T2D complications, Sepecially NAFLD. This work is critically urgent as the U.S. burden of NAFLD is rising, and several drugs for NAFLD in T2D will come to market soon; this proposal will support equitable use of current and emerging therapies for NAFLD, assuring that those with the greatest need are able to access effective treatment. Because current services are already struggling to reach rising numbers of patients with NAFLD, a major strength of this proposal is its support of multidisciplinary efforts to tackle this public health threat.

<u>Innovation</u>: This proposal is novel in multiple ways. First, the drivers underlying health disparities in NAFLD detection are poorly understood, and this proposal will address this gap. Second, there are no existing interventions to promote detection and management of NAFLD as part of T2D care, and certainly none to address disparities in these areas. Third, I am proposing an innovative intervention development approach that will leverage community engagement resources at Duke and maximize intervention relevance and feasibility through use of stakeholder input. No studies have queried minority communities to understand how best to design/deliver an intervention to improve outcomes in NAFLD and T2D. Notably, this proposal will proactively improve the care of an exceedingly high-risk, high-cost group through a joint **T2D/NAFLD intervention**. To our knowledge, this will be the first intervention geared towards intensively co-managing these linked conditions.

#### Research Strategy/Approach

This project will assess the feasibility and acceptability of an intervention for improved detection and evidence-based care of NAFLD in Latinx and Black patients with T2D.

PI: Anastasia-Stefania Alexopoulos, MD

Version 2: May 31, 2024


Rationale: Below is a conceptual framework that has guided the design, and will inform the execution, of our intervention. This framework includes features of the Health Belief Model (HBM)<sup>14</sup> to highlight patient-level strategies for disease prevention, and the Chronic Care Model (CCM)<sup>15</sup> to highlight the system-level components aimed at improving the care of NAFLD. As depicted in the Figure below, this intervention represents an innovative approach to *redesigning care* and using available *EHR* to promote equitable detection of NAFLD (right side of figure). Once detected, we will engage patients with NAFLD and T2D in strategies to promote their overall health and halt, or even reverse their NAFLD. These patient-level approaches will consider how to alter patient perceptions (i.e., *perceived threat* of NAFLD, *perceived benefits & barriers*) and understand patient *cues to action*, to promote patient engagement with the care plan (left side of Figure). The ultimate objective of this project is to lead to *productive interactions* between patients and the care teams (center of Figure) that will ultimately lead to better detection and care of NAFLD in those at highest risk. Prior work has helped us develop this intervention in a culturally-appropriate manner to allow us to reach high-risk racial/ethnic groups with T2D and NAFLD. This will be a feasibility pilot.

Figure: Conceptual framework guiding intervention design and execution Underdiagnosis of NAFLD and complications in T2D Insufficient use of evidence-based T2D therapies Disparities in NAFLD outcomes KL2 intervention Perceived threat of Clinical information **NAFLD** systems (EHR) Prepared, Informed. Productive Perceived benefits Proactive Activated patient-provider & barriers Care team interactions patient Delivery system redesign Cues to action Improved NAFLD diagnosis earlier in course High utilization of evidence-based T2D therapies Equity in detection & care of NAFLD in T2D

PI: Anastasia-Stefania Alexopoulos, MD

Version 2: May 31, 2024


Intervention content and design: The first intervention component will involve proactive detection of NAFLD in Latinx/Black patients with T2D using DEDUCE; this EHR-based approach will allow us to identify eligible study participants in DUHS based on our inclusion/exclusion criteria listed below. The next intervention component will focus on delivery of evidence-based care, which will rely on a proactive care team that is knowledgeable about NAFLD and can intervene, as well as an informed and activated patient who wants to engage with care.

Once identified, patients will receive the following guideline-concordant content as part of the intervention: a) diet/lifestyle support, with counseling on hypocaloric diet and moderate-intensity exercise;<sup>5</sup> b) NAFLD education;<sup>5</sup> c) medication management, with proactive use of T2D medications known to be protective against NAFLD progression (pioglitazone, GLP-1RA, SGLT2i);<sup>5, 7, 16</sup> and d) clinically-indicated liver testing and care based on guidelines.<sup>5</sup> The content of this intervention will be delivered remotely via telehealth approaches. In order to ensure feasibility within the proposed KL2 timeline, we have limited the pilot duration to 3 months. This will allow time to observe change in liver enzymes, as well as HbA1c. Table 1

shows when intervention content will be delivered throughout the

<u>Study population:</u> We will enroll 10-15 Latinx/Hispanic and 10-15 Black patients with T2D and NAFLD, based on elevated ALT and exclusion of other liver diseases (e.g., viral hepatitis, alcohol abuse).

#### Research activity:

**Detection of NAFLD in T2D**: The Duke DEDUCE tool will be used to generate a report of potentially eligible Latinx and Black patients with an ICD code for T2D (E11.xx) and at least one ALT >40 IU/mL in males or > 31 IU/mL in females<sup>17</sup> in the preceding 12 months. For this feasibility pilot, we will also restrict eligibility to patients who have a PCP or Endocrinologist in DUHS to facilitate communication regarding T2D medication changes during the study period. We anticipate >2,000 patient will meet our inclusion and exclusion criteria. A report will be exported from DEDUCE and I will review the charts of potentially eligible patients to exclude individuals with liver dysfunction likely due to an etiology other than NAFLD. We will not exclude patients with an ICD-10 code for NASH (K75.81), as long as they are not medically optimized (i.e. on pioglitazone and GLP-1RA), since these individuals serve to benefit from the intervention.

The first 50 patients who meet eligibility will be mailed a letter or sent a MyChart message with opt-out instructions. Patients who do not opt out will be contacted by phone and, if interested, they will sign an e-

consent form via REDCap. In parallel to the above recruitment approach, we will also advertise this study in the community with the help of community partners that had assisted us in the design of the intervention, i.e., Latin-19 group and the AME Zion partnership. An IRB-approved flyer (with brief inclusion/exclusion criteria) will be created and placed in community spaces with the help of our community partners. Community members who are interested in the study, and who

| Table 1: NAFLD-DM study visits and timing | Months | | | |
|-----------------------------------------------------|--------|---|---|---|
| • | 0 | 1 | 2 | 3 |
| Enrollment, consent review (~20 min, remote visit) | Х | | | |
| Surveys (~20-30 min, online or on phone) | Х | | | Х |
| NAFLD education (~30 min, remotely) | Х | | | |
| Diet and lifestyle support (~30 min each, remotely) | Х | Х | Х | |
| Medication changes (~20 min, remotely) * | 0 | 0 | 0 | 0 |
| If indicated, ordering tests and referrals * | 0 | 0 | 0 | 0 |
| Interviews (~30 min, remotely) | | | | Х |
| Interviews (~30 min, remotely) | -1 | | | |

<sup>\*</sup>Timing of med changes and ordering of tests/referrals will vary by participant.

are also part of DUHS, will be provided with a study contact number to let us know of their interest. We will use the EHR to determine their eligibility, and if eligible, consent will be obtained as above.

Baseline surveys will be conducted by phone or completed online via Duke REDCap. For participants completing surveys by phone, we will ensure that a copy of the survey is mailed or emailed in advance, in case participants prefer to review content in advance. We will survey: self-efficacy,<sup>18</sup> and quality of life surveys<sup>19</sup>). The most recent BMI in the EHR will be used for the purpose of characterizing the participant population – if there is no BMI documented within 1 year of enrollment, we will count BMI data as missing. For HbA1c, if there is no documented HbA1c within 3 months of enrollment to the study, or ALT and ALT within 6 months of enrollment, we will order these tests to be completed at baseline.

x Visits that will occur for all participants.

o Visits that may or may not occur and are dependent upon individual needs.

PI: Anastasia-Stefania Alexopoulos, MD

Version 2: May 31, 2024


**Evidence-based care of NAFLD in T2D:** Intervention content will include: 1) NAFLD education; 2) diet/lifestyle support; 3) T2D medication management; and 4) clinically-indicated liver testing and care. Dr. Alexopoulos (PI) and the Clinical Research Coordinator (CRC) will deliver NAFLD education and diet/lifestyle support content. Dr. Alexopoulos (PI) will conduct medication management, which will involve review of glycemic trends, assessment of hypoglycemia and adjustment of the T2D regimen to accommodate initiation of pioglitazone, GLP-1RA and/or SGLT2i. The order in which these medications are considered will depend on clinical judgement, patient preference and cost, but GLP-1RA will be prioritized as appropriate, since this class has potent weight loss effects. Also, at baseline (and as indicated throughout the study), Dr. Alexopoulos (PI) will review clinical data and order clinically-indicated liver testing based on guidelines. Surveys and clinical evaluation will be repeated at study conclusion. A treatment acceptability measure (TAP) will be administered at conclusion to gauge intervention acceptability. A detailed summary of data collection and outcome measures can be seen in Table 3.

| Table 3: Detailed summary of data collection and outcomes | Method | Timing |
|---|---|---|
| | y outcomes | |
| Feasibility | | |
| System-level NAFLD detection | Patients who met criteria for NAFLD after chart review / total number of potentially-eligible patients based on our EHR criteria | 3 months |
| Recruitment rate* | Patients eligible and sent letter or<br>MyChart message / Patients<br>enrolled | 3 months |
| Retention rate | Patients enrolled / Patients completed study | 3 months |
| Visit completion rate | Total study visits completed / total study visits scheduled | 3 months |
| Acceptability | | |
| | TAP measure <sup>20</sup> | 3 months |
| | Qualitative interviews | 3 months |
| Secondary ou | tcomes of interest | |
| Medication changes made during the study | Study visit notes in EHR | 0, 3 months |
| Proportion of patients in whom clinically-<br>indicated tests were ordered (e.g. labs, referral,<br>imaging). | Study visit notes in HER | 0, 3 months |
| Psychosocial constructs Self-efficacy Autonomy support Quality of life | 6-item SEMCD <sup>21</sup><br>HCCQ Diabetes <sup>18</sup><br>SF-12 <sup>19</sup> | 0,3 months |
| | characterize population | |
| Social and demographic Age, sex, race/ethnicity, marital status, education, employment, tobacco use, alcohol use, SDOH screen (food insecurity, housing instability, lack of transportation) | Self-reported surveys | 0 months |
| Health literacy/numeracy | NVS | 0 months |
| Medication adherence | VMNQ <sup>22</sup> | 0 months |
| Clinical Baseline knowledge of NAFLD, years with diabetes, medical history, medication use | Self-reported surveys | 0 months |

PI: Anastasia-Stefania Alexopoulos, MD Page **5** of **7** 

Version 2: May 31, 2024

| Labs: HbA1c, AST, ALT | Use from EHR if collected within 3 months of baseline visit. Otherwise, research labs collected in DUHS at specified time points. | 0 months |
|---|---|---|
| Biomedical<br>Height, weight, BMI | From EHR (last recorded values) | 0 months |

<sup>\*</sup>We will also track the number of participants who expressed interest in the study based on our recruitment flyer, and examine the recruitment rate via this approach (i.e., patients who expressed interest / patients enrolled. **Abbreviations**: TAP=Treatment Acceptability & Preferences; SDOH=social determinates of health; NAFLD=nonalcoholic fatty liver disease; BMI=body mass index; HER=electronic health record; SEMCD=Self-efficacy to Manage Chronic Disease Scale; VMNQ=Voils Medication Non-Adherence Questionnaire; NVS=Newest Vital Sign; HCCQ=Healthcare Climate Questionnaire.

**Participant interviews**: At study conclusion, individual 30-minute virtual interviews will be conducted with all study participants. The primary purpose will be to assess intervention acceptability and to gain specific feedback about intervention content. Thematic saturation is expected by 12 interviews.<sup>22</sup>

<u>Quantitative analysis:</u> Intervention feasibility will be evaluated by examining recruitment rates, retention rates, and study visit completion rates. For the TAP measure, mean score and standard deviation will be calculated. This feasibility pilot will not be powered to examine changes in clinical measures (e.g., HbA1c, ALT).

<u>Qualitative analysis:</u> All interviews will be digitally recorded and transcribed. Transcripts will be analyzed with direct content analysis.<sup>23</sup>

PI: Anastasia-Stefania Alexopoulos, MD Page **6** of **7** 

Version 2: May 31, 2024

#### References

- 1. Younossi ZM, Stepanova M, Rafiq N, et al. Nonalcoholic steatofibrosis independently predicts mortality in nonalcoholic fatty liver disease. *Hepatol Commun*. Jul 2017;1(5):421-428. doi:10.1002/hep4.1054
- 2. Diabetes Mellitus. Federal Practitioner. 2017;
- 3. Samji NS, Snell PD, Singal AK, Satapathy SK. Racial Disparities in Diagnosis and Prognosis of Nonalcoholic Fatty Liver Disease. *Clin Liver Dis* (Hoboken). Aug 2020;16(2):66-72. doi:10.1002/cld.948
- 4. Alexopoulos AS, Crowley MJ, Wang Y, et al. Glycemic Control Predicts Severity of Hepatocyte Ballooning and Hepatic Fibrosis in Nonalcoholic Fatty Liver Disease. *Hepatology*. Mar 16 2021;doi:10.1002/hep.31806
- 5. Chalasani N, Younossi Z, Lavine JE, et al. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. *Hepatology*. Jan 2018;67(1):328-357. doi:10.1002/hep.29367
- 6. American Diabetes A. 4. Comprehensive Medical Evaluation and Assessment of Comorbidities: Standards of Medical Care in Diabetes-2021. *Diabetes Care*. Jan 2021;44(Suppl 1):S40-S52. doi:10.2337/dc21-S004
- 7. Newsome PN, Buchholtz K, Cusi K, et al. A Placebo-Controlled Trial of Subcutaneous Semaglutide in Nonalcoholic Steatohepatitis. *N Engl J Med*. Mar 25 2021;384(12):1113-1124. doi:10.1056/NEJMoa2028395
- 8. Raj H, Durgia H, Palui R, et al. SGLT-2 inhibitors in non-alcoholic fatty liver disease patients with type 2 diabetes mellitus: A systematic review. *World J Diabetes*. Feb 15 2019;10(2):114-132. doi:10.4239/wjd.v10.i2.114
- 9. Alexopoulos AS, Duffy R, Kobe EA, et al. Underrecognition of nonalcoholic fatty liver disease in poorly-controlled diabetes: A call to action in diabetes care. *J Endocr Soc (In Press)*. 2021;
- 10. Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. *Hepatology*. Jan 2018;67(1):123-133. doi:10.1002/hep.29466
- 11. Shetty A, Syn WK. Health and Economic Burden of Nonalcoholic Fatty Liver Disease in the United States and Its Impact on Veterans. *Fed Pract*. Jan 2019;36(1):14-19.
- 12. Younossi ZM, Blissett D, Blissett R, et al. The economic and clinical burden of nonalcoholic fatty liver disease in the United States and Europe. *Hepatology*. Nov 2016;64(5):1577-1586. doi:10.1002/hep.28785
- 13. Haw JS, Shah M, Turbow S, Egeolu M, Umpierrez G. Diabetes Complications in Racial and Ethnic Minority Populations in the USA. *Curr Diab Rep.* Jan 9 2021;21(1):2. doi:10.1007/s11892-020-01369-x
- 14. MH B. The Health Belief Model and personal health behavior. *Health Education Monographs*. 1974;2:324–508.
- 15. EH W. Chronic disease management: What will it take to improve care for chronic illness? *Effective Clinical Practice*. 1998;1(1):2-4.
- 16. American Diabetes A. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2021. *Diabetes Care*. Jan 2021;44(Suppl 1):S111-S124. doi:10.2337/dc21-S009
- 17. Kanwal F, Kramer JR, Mapakshi S, et al. Risk of Hepatocellular Cancer in Patients With Non-Alcoholic Fatty Liver Disease. *Gastroenterology*. Dec 2018;155(6):1828-1837 e2. doi:10.1053/j.gastro.2018.08.024
- 18. Williams GC, Freedman ZR, Deci EL. Supporting autonomy to motivate patients with diabetes for glucose control. *Diabetes Care*. Oct 1998;21(10):1644-51. doi:10.2337/diacare.21.10.1644
- 19. Ware J, Jr., Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. *Med Care*. Mar 1996;34(3):220-33. doi:10.1097/00005650-199603000-00003
- 20. Sidani S, Epstein DR, Bootzin RR, Moritz P, Miranda J. Assessment of preferences for treatment: validation of a measure. *Res Nurs Health*. Aug 2009;32(4):419-31. doi:10.1002/nur.20329
- 21. Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. *J Clin Epidemiol*. Nov 2014;67(11):1265-73. doi:10.1016/j.jclinepi.2014.06.009
- 22. G. G. A. B, Johnson L. How Many Interviews Are Enough?: An Experiment with Data Saturation and Variability. *Field Methods*. 2006;18(1):59-82.
- 23. Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. *Qual Health Res.* Nov 2005;15(9):1277-88. doi:10.1177/1049732305276687

PI: Anastasia-Stefania Alexopoulos, MD

Version 2: May 31, 2024
